CLINICAL TRIAL: NCT02742961
Title: Impact of Peripheral Nerve Blockade on Outcomes After Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dan McIsaac, Associate Scientist, Ottawa Hospital Research Institute
Other Study IDs: DM1
Record Dates: First submitted 2016-04-13; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Pain; Osteoarthritis
Keywords: orthopedics; anesthesiology; nerve block; length of stay; Patient readmission
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Peripheral nerve block: Intervention arm. Participants who receive a peripheral nerve block identified through submission of an appropriate physician billing code
  Interventions: Other: Peripheral nerve block
- No peripheral nerve block: Control arm. Participants who do not receive a peripheral nerve block identified through lack of a submission of an appropriate physician billing code

INTERVENTIONS:
Other: Peripheral nerve block — A physician billing code for deposition of a local anesthetic solution around an anatomically defined nerve or nerve plexus
  Groups: Peripheral nerve block

SUMMARY:
Pain is common after knee replacement surgery and can impact a variety of patient outcomes. Peripheral nerve blocks provide improved pain control and may improve function. However, their impact on other outcomes is poorly described. Therefore, this comparative effectiveness study will estimate the independent association between nerve blocks and health outcomes after knee replacement surgery.

DETAILED DESCRIPTION:
This retrospective, population-based cohort study will evaluate the comparative effectiveness of peripheral nerve blocks on patient and health system outcomes after elective total knee replacement surgery.

The investigators will develop a non-parsimonious propensity score to control for potential indication bias and confounding in this observational study. Using the propensity score the investigators will match patients who receive a peripheral nerve block to a patient who did not to estimate the independent association of peripheral nerve blocks with our study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* first primary total knee replacement during the study period

Exclusion Criteria:

* Revision arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults having their first total knee replacement during the study period
Sampling Method: Non-Probability Sample
Enrollment: 178214 (Actual)
Dates: Start 2002-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Day of surgery to day of discharge, or up to 365 days, whichever comes first
  Determined from the Canadian Institute for Health Information Discharge Abstract Database record for the index hospitalization

SECONDARY OUTCOMES:
Hospital readmission | The outcome ascertainment window starts on the day of discharge and extends up to 30 days after surgery. Any readmission in this time period will be considered an event.
  Determined from the Canadian Institute for Health Information Discharge Abstract Database through identification of a new record after discharge from the index hospitalization
In-hospital fall | hospital admission
  Determined using validated International Classification of Diseases Tenth edition codes for falls from the index hospitalization Discharge Abstract Database record
Emergency department visit | The outcome ascertainment window starts on the day of discharge and extends up to 30 days after surgery. Any emergency department visit in this time period will be considered an event.
  Defined as the creation of a record in the National Ambulatory Care Reporting System for an emergency department visit that occurs after discharge and before 30 days after discharge

OTHER OUTCOMES:
All cause mortality | Day of surgery to 30 days after surgery
  Identified from the Registered Person's Database that records the date of death for all residents of Ontario

CONTACTS AND LOCATIONS:
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No